CLINICAL TRIAL: NCT07024147
Title: An Open-Label, Single-arm Study of JWCAR239 in the Treatment of Relapse / Refractory (R/R) B Cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: JWCAR239 in Patients With B Cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Shanghai JW Therapeutics Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR239001
Record Dates: First submitted 2025-05-27; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Large B Cell Diffuse Lymphoma; Follicular Lymphoma; Marginal Zone B Cell Lymphoma; Mantle Cell Lymphoma (MCL)
Keywords: CAR-T; dual target; B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR239 arm (Experimental): Participants will receive cyclophosphamide 250-300mg/m^2/day intravenously (IV) and fludarabine 25-30mg/m^2/day IV conditioning chemotherapy for 3 days followed by JWCAR239 administered as a single IV infusion at a target dose of 2 .5-30x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells on Day 1.
  Interventions: Biological: JWCAR239; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: JWCAR239 — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells targeting CD19/CD20
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
JWCAR239 is a CD19/CD20 CAR-T product. This trial is intended to evaluate the safety, PK/PD and efficacy of JWCAR239 in patients with B Cell Non-Hodgkin Lymphoma (B-NHL)

DETAILED DESCRIPTION:
JWCAR239 is a CD19/CD20 CAR-T product. By targeting both CD19 and CD20, it is expected to overcome some limitations with CD19 or CD20 single target products. In this study, patients with B B-NHL will be enrolled to receive JWCAR239. PK/PD properties and preliminary efficacy and safety will be evaluated. Each subject will receive JWCAR239 once and is followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed B-NHL with immunohistochemical positivity for CD20 and/or CD19 (accepting previous pathological reports and/or pathological review results of previous or fresh tumor tissues). According to the 2022 World Health Organization (WHO) classification, the pathological types include:Diffuse large B-cell lymphoma, Follicular large B-cell lymphoma (FL3B),Large B-cell lymphoma transformed from indolent B-NHL, Follicular lymphoma (excluding in situ follicular lymphoma, pediatric-type follicular lymphoma, and duodenal-type follicular lymphoma),Marginal zone lymphoma Mantle cell lymphoma (excluding in situ mantle cell neoplasms and leukemic non-nodal mantle cell lymphoma)
2. Relapsed or refractory disease after receiving two or more lines of adequate treatment, or failure after autologous hematopoietic stem cell transplantation (ASCT).
3. CT-measurable lesions and PET-evaluable positive lesions as defined by the 2014 Lugano criteria (lymph node or extranodal lesions must have two measurable diameters; lymph node lesions must have a long diameter >1.5 cm, and extranodal lesions must have a long diameter >1 cm).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ function:

   Sufficient bone marrow function as assessed by the investigator (absolute neutrophil count ≥1,000/μL after at least 72 hours off growth factors; platelet count ≥50,000/μL without blood transfusion within 7 days; absolute lymphocyte count ≥100/μL).

   Serum creatinine ≤1.5× upper limit of normal (ULN) or creatinine clearance ≥50 mL/min (calculated by the Cockcroft-Gault formula).

   Alanine aminotransferase (ALT) ≤5×ULN and total bilirubin <2×ULN (or <3×ULN for subjects with Gilbert syndrome or hepatic involvement by lymphoma).

   Pulmonary function: ≤ CTCAE Grade 1 dyspnea and SpO2 ≥92% in room air. Cardiac function: Left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiography.
6. Adequate vascular access for leukapheresis.
7. Expected survival >12 weeks.
8. Non-abstinent female subjects of childbearing potential must agree to use a highly effective contraceptive method plus an additional barrier method from at least 28 days before lymphodepletion until 2 years after JWCAR239 infusion. Male subjects with fertile partners must agree to use effective contraception from at least 28 days before lymphodepletion until 2 years after JWCAR239 infusion and must not donate semen or sperm throughout the study.

Exclusion Criteria:

1. Lymphoma involving the central nervous system (CNS).
2. EBV-positive DLBCL or Richter transformation of chronic lymphocytic leukemia.
3. History of other malignant tumors with complete remission for less than 2 years, or current presence of other malignant tumors (exceptions to the 2-year restriction include: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, treated localized prostate cancer, biopsy-confirmed cervical in situ carcinoma, or cervical smears showing squamous intraepithelial lesions, or completely resected tumors with low recurrence potential as assessed by the investigator).
4. At screening, the subject has:

   Active hepatitis B or C (subjects with HBV DNA or HCV RNA below the lower limit of the central reference value by PCR may be enrolled). For occult or prior HBV-infected subjects, prophylactic antiviral therapy and regular monitoring of HBV-DNA are required.

   Human immunodeficiency virus (HIV) infection or syphilis infection.
5. Acute deep vein thrombosis (DVT) (tumor thrombus or thrombus) or pulmonary embolism (PE) within 3 months prior to informed consent signing.
6. Receiving anticoagulant therapy for acute DVT or PE within 3 months prior to informed consent signing (prophylactic treatment ).
7. Uncontrolled systemic fungal, bacterial, viral, or other infections.
8. Acute or chronic graft-versus-host disease (GvHD).
9. History of any of the following cardiovascular diseases within the past 6 months: New York Heart Association (NYHA) Class III or IV heart failure, coronary angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart diseases.
10. Clinically significant CNS disease or symptoms at screening or within the past 6 months, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychiatric disorders.
11. Pregnant or lactating women. Females of childbearing potential must have a negative serum pregnancy test within 48 hours before starting lymphodepletion chemotherapy.
12. Use of any of the following drugs or treatments within the specified time before leukapheresis:

    Alemtuzumab within 6 months before leukapheresis. Bendamustine within 6 months before leukapheresis. Cladribine within 3 months before leukapheresis. Fludarabine within 3 months before leukapheresis. Anti-CD20 monoclonal antibodies within 7 days before leukapheresis. Venetoclax within 4 days before leukapheresis. Idelalisib within 2 days before leukapheresis. Lenalidomide within 1 day before leukapheresis. Pharmacological doses of corticosteroids (defined as prednisone >5 mg/day or equivalent) within 7 days before leukapheresis or within 72 hours before JWCAR239 injection. Physiological replacement, topical, and inhaled steroids are permitted.

    Chemotherapy (e.g., vincristine, rituximab, cyclophosphamide) required to control the disease after leukapheresis must have been discontinued ≥7 days before lymphodepletion chemotherapy.

    Administration of non-lymphocyte-toxic cytotoxic chemotherapy within 1 week before leukapheresis. Enrollment is permitted if the oral chemotherapy has undergone at least 3 half-lives before leukapheresis.

    Receipt of lymphocyte-toxic chemotherapy (e.g., cyclophosphamide, ifosfamide, chlorambucil, or melphalan) within 2 weeks before leukapheresis.

    Use of investigational drugs within 4 weeks before leukapheresis. However, enrollment is permitted if the investigational treatment was ineffective or caused disease progression, and at least 3 half-lives have elapsed before leukapheresis.

    Treatment with immunosuppressive agents (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutic drugs, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL-6, or anti-IL-6R) within 4 weeks before leukapheresis and JWCAR239 injection.

    Receipt of donor lymphocyte infusion (DLI) within 6 weeks before JWCAR239 injection.

    Radiation therapy involving large bone marrow areas (e.g., sternum or pelvis) within 6 weeks before leukapheresis. Subjects are eligible only if the disease progresses at the radiation site or PET-positive lesions exist in non-irradiated areas. If PET-positive lesions exist in non-irradiated areas, radiation therapy to a single lesion is permitted within 2 weeks before leukapheresis.
13. Any other significant disease, abnormality, or condition that, in the investigator's judgment, renders the subject unsuitable for participation in the study or places the subject at risk. Any factors affecting compliance with the protocol, including uncontrollable medical, psychological, family, sociological, or geographical factors; or unwillingness or inability to adhere to the procedures required by the study protocol.
14. Prior allogeneic hematopoietic stem cell transplantation.
15. Prior treatment with CAR+ T cells or other genetically modified T cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The rate of Dose Limiting Toxicity events | 28 days
  Dose-Limiting Toxicity (DLT) refers to a specific type of adverse effect or toxic reaction caused by a drug or treatment that is severe enough to prevent an increase in dose or continuation of treatment.
AE and SAE rate | up to 2 years
  ny adverse event (AE) or serious adverse event (SAE) occurring after JWCAR239 administration

SECONDARY OUTCOMES:
Pharmacokinetic (PK)- Cmax of JWCAR239 | from baseline up to 2 years
  Maximum observed concentration of JWCAR239 in peripheral blood
PD | from baseline up to 2 years
  Peripheral blood levels of CD19+ and/or CD20+ B cells
overall response rate (ORR) | from baseline up to 2 years
  ORR is the proportion of subjects who achieve positive response to the treatment. It includes complete response and partial response.
complete response rate (CRR) | from baseline up to 2 years
  CRR refers to the proportion of subjects whose cancer signs disappear
duration of response(DOR) | from baseline up to 2 years
  in subjects with hematology malignancy The duration of a subject staying in response state
progression free survival(PFS) | from baseline up to 2 years
  the length of time during and after treatment that a subject lives with the disease without the disease worsening or progressing
Overall survival(OS) | from baseline up to 2 years
  the length of time from the start of treatment that patients are still alive
Pharmacokinetic (PK)- Tmax of JWCAR239 | up to 2 year after JWCAR239 infusion
  Time to maximum concentration of JWCAR239 in the peripheral blood
Pharmacokinetic (PK)- AUC of JWCAR239 | up to 2 year after JWCAR239 infusion
  Area under the concentration vs time curve of JWCAR239

OTHER OUTCOMES:
The change of serum cytokines concentration | from baseline up to 2 years
  The change of serum cytokines concentration after JWCAR239 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No